CLINICAL TRIAL: NCT07023796
Title: Comparison of the Efficacy Between Autologous Fat Infiltration and Treatment With General Measures in the Management of Radiotherapy-induced Radiodermatitis in Breast Cancer Patients.
Brief Title: Autologous Fat Infiltration Versus General Measures as Treatment in Radiodermatitis Induced for Radiotherapy in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Clotilde Fuentes-Orozco, Principal investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2023-1301-147
Record Dates: First submitted 2025-06-04; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Radio Dermatitis; Radiotherapy
Keywords: Autologus Fat Filtration; Radiodermatitis; Breast cancer; Nanofat
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who received general care (No Intervention): Patients who received daily skin washing with warm water and mild soap (pH neutral, fragrance free) without scrubbing.
- Patients who received autologous fat filtration (Active Comparator): Patients who underwent a surgical procedure and autologous fat processing for subsequent fat filtration.
  Interventions: Procedure: Autologous fat filtration

INTERVENTIONS:
Procedure: Autologous fat filtration — Patients who underwent a surgical procedure and autologous fat processing for subsequent fat filtration.
  Arms: Patients who received autologous fat filtration

SUMMARY:
Radiodermatitis is a major problem in oncologic patients, fat grafts previously used for cosmetic procedures have been shown to have regenerative power due to their stem cell content. Our purpose was to compare the clinical changes in the treatment of radiation dermatitis in breast cancer patients with the application of fat graft versus traditional therapy with general measures.A randomized controlled clinical trial was performed, 22 patients were recruited and randomly assigned to one of two groups: an intervention group that received an autologous fat graft and a control group that received treatment with general measures; a 6-week follow-up was performed to determine the presence and classification of radiodermatitis using the LENT/SOMA scales, as well as biopsies. Women were included, with a diagnosis of breast cancer, Eastern Cooperative Oncology Group 0 or 1, attended in our hospital during September 2023 to October 2024, older than 18 years, undergoing lumpectomy or mastectomy and in radiotherapy as part of the treatment scheme for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with a confirmed diagnosis of common bile duct cyst by imaging studies and/or intraoperative findings.
* Patients who received surgical treatment at the institution during the study period.
* Clinical records with complete information for analysis.

Exclusion Criteria:

* Patients who do not consent to their inclusion in the study or who for any physical or mental reason are unable to give their consent (patients with cognitive impairment, etc.).
* Pediatric patients (<18 years).
* Incomplete clinical records or with loss of postoperative follow-up.
* Patients with diagnosis of other biliary pathology without evidence of common bile duct cyst.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with radiodermatitis | From the start to six week later
  The number of patients with radiodermatitis secondary to radiotherapy will be measured from the day they received the treatment until six weeks later.

CONTACTS AND LOCATIONS:
Locations (1):
- Belisario Dominguez 1000, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No